CLINICAL TRIAL: NCT00910169
Title: Evaluation of Hospitalization for Anorexia Nervosa: Efficacy of Treatment and Predictive Factors of Outcome.
Brief Title: Evaluation of Hospitalization for Anorexia Nervosa (EVALuation de l'Apport de l'HOSPITalisation Pour Anorexie Mentale : EVALHOSPITAM)
Acronym: EVHAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Ministry of Health, France (Other Government); National Research Agency, France (Other); National Health Insurance Fund (Other); Fondation de la Mutuelle Générale de l'Education Nationale (Unknown); Fondation de France (Other)
Responsible Party: Nathalie Godart, M.D., Ph.D., Institut Mutualiste Montsouris
Other Study IDs: Eudract: 2007 -A01110-53; ANR-0-JC0719-6328; PHRC AOM 06 020
Record Dates: First submitted 2009-05-26; First posted 2009-05-29 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2009-05

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; treatment; inpatient; efficacy; outcome
MeSH Terms: conditions — Anorexia Nervosa | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — all biological analysis during hospitalisation, serotonin , tryptophan, CD4/CD8
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- inpatient treatment: naturalistic treatment no modification: observational study
  Interventions: Other: inpatient treatment

INTERVENTIONS:
Other: inpatient treatment — Hospitalisation modalities are described but are naturalistic
  Other Names: naturalistic treatment

SUMMARY:
The objective of this research is to evaluate the efficacy of five different in-patient treatment modalities and predictive factors of outcome for anorexia nervosa. The primary hypothesis is that the different treatment types impact outcome of patients at discharge from inpatient treatment and at one year follow-up, even after adjustment for confounding factors (age, length of illness, number of previous hospitalizations, clinical state at intake).

DETAILED DESCRIPTION:
This study will evaluate global, psychiatric, somatic and psychosocial outcome for inpatients with anorexia nervosa through three evaluations (intake, discharge and one-year follow-up). The study will also consider five types of in-patient treatment in a naturalistic setting (i.e., patients will not be assigned to different treatment conditions; rather, we will study inpatient care as it exists today). The five treatment modalities to be studied are:

1. Discharge weight objectives.
2. The practice of a separation period.
3. The use of clear nutritional and dietary objectives (cognitive/behavioural).
4. The intensity of family involvement in treatment.
5. Stabilisation phase before ending inpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients who accept participation between 8 and 50 years old, consecutively hospitalized for a DSM IV diagnosis of Anorexia Nervosa in one of the departments participating in this research by necessity of physical condition (BMI < 15, rapid weight loss) or psychological condition
* Parents of participating patients still living with their parents who accept participation

Exclusion Criteria:

* Refusal of research
* Patients who do not speak French
* Patients with a related somatic illness (diabetes, Crohn's disease, metabolic illness)
* Patients not covered by social security health insurance

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalisied in 11 tertiary centers for eating disorders in france
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Morgan and Russell score | one year follow-up

SECONDARY OUTCOMES:
Nutritional status | one year follow-up
Eating disorders symptoms and diagnosis | one year follow-up
Psychiatric symptoms and disorders | one year follow-up
Cognitive functioning | one year follow-up
Somatic symptoms and complications | one year follow-up
Social adjustment | one year follow-up
Quality of life | one year follow-up
Family relationships | one year follow-up
Re-hospitalization | one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Godart Nathalie, PhD, Principal Investigator — INSERM and Institut Mutualiste Montsouris
Locations (1):
- Insitut Mutualiste Montsouris, Paris, France

REFERENCES:
- [Derived] Duclos J, Piva G, Riquin E, Lalanne C, Meilleur D, Blondin S; EVHAN Group; Cook-Darzens S, Godart N. Caregivers in anorexia nervosa: is grief underlying parental burden? Eat Weight Disord. 2023 Feb 20;28(1):16. doi: 10.1007/s40519-023-01530-x. PMID 36807834